CLINICAL TRIAL: NCT01408576
Title: A Phase 3, Multicenter, Open-label, Extension Study to Assess the Safety and Tolerability of Epratuzumab Treatment in Systemic Lupus Erythematosus Subjects
Brief Title: Open Label Extension Study of Epratuzumab in Subjects With Systemic Lupus Erythematosus
Acronym: EMBODY4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL0012; 2010-020859-30 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2016-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-Cell immunotherapy; Epratuzumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epratuzumab 600 mg per week (Experimental): 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
  Interventions: Drug: Epratuzumab
- Epratuzumab 1200 mg every other week (Experimental): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over sixteen 12 week treatment cycles
  Interventions: Drug: Epratuzumab

INTERVENTIONS:
Drug: Epratuzumab — 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over eight 12-week treatment cycles
  Arms: Epratuzumab 600 mg per week
Drug: Epratuzumab — 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over eight 12 week treatment cycles
  Arms: Epratuzumab 1200 mg every other week

SUMMARY:
The primary objective of the study is assess the safety and tolerability of long-term epratuzumab treatment in subjects with Systemic Lupus Erythematosus (SLE)

DETAILED DESCRIPTION:
Treatment period was extended by 2 years to a total of 4 years and an amendment was prepared accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the double-blind study SL0009 (NCT01262365) or SL0010 (NCT01261793) or terminated prematurely at Week 16 or later in SL0009 or SL0010 due to lack of efficacy and would, in the opinion of the investigator, continue to benefit from continued epratuzumab treatment
* Subject has completed open-label study SL0006 (NCT00383513) or SL0008 (NCT00660881), and would, in the opinion of the investigator, continue to benefit from continued epratuzumab treatment
* Women of childbearing potential must agree to use an acceptable method of birth control

Exclusion Criteria:

* Subjects with active, severe, neuropsychiatric SLE, defined as any neuropsychiatric element scoring British Isles Lupus Assessment Group Index (BILAG) level A disease
* Subjects with active, severe SLE disease activity which involves the renal system
* Subjects with concurrent relevant medical conditions like defined chronic infections or high risk of new significant infections
* Substance abuse or dependence
* History of malignant cancer
* Subjects with any other condition which, in the investigator's judgment, would make the subject unsuitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (228):
- United States (78):
  - 539, Birmingham, Alabama
  - 557, Little Rock, Arkansas
  - 515, Hemet, California
  - 544, Huntington Beach, California
  - 550, La Jolla, California
  - 031, Los Angeles, California
  - 051, Los Angeles, California
  - 089, Los Angeles, California
  - 531, San Leandro, California
  - 594, Thousand Oaks, California
  - 558, Torrance, California
  - 048, Aurora, Colorado
  - 037, Colorado Springs, Colorado
  - 532, Denver, Colorado
  - 511, Bridgeport, Connecticut
  - 039, Farmington, Connecticut
  - 042, Aventura, Florida
  - 514, Brandon, Florida
  - 090, Clearwater, Florida
  - 092, DeBary, Florida
  - 533, Fort Lauderdale, Florida
  - 064, Jupiter, Florida
  - 070, Ormond Beach, Florida
  - 084, Palm Harbor, Florida
  - 518, Plantation, Florida
  - 585, Port Orange, Florida
  - 050, Tampa, Florida
  - 538, Tampa, Florida
  - 087, Vero Beach, Florida
  - 537, Atlanta, Georgia
  - 044, Duluth, Georgia
  - 590, Idaho Falls, Idaho
  - 052, Chicago, Illinois
  - 096, Indianapolis, Indiana
  - 060, Shreveport, Louisiana
  - 513, Lansing, Michigan
  - 599, Lansing, Michigan
  - 047, Saint Clair Shores, Michigan
  - 575, Florissant, Missouri
  - 549, St Louis, Missouri
  - 596, Nashua, New Hampshire
  - 568, Freehold, New Jersey
  - 593, Trenton, New Jersey
  - 067, Las Cruces, New Mexico
  - 551, Brooklyn, New York
  - 553, Great Neck, New York
  - 545, Manhasset, New York
  - 053, New York, New York
  - 577, Roslyn, New York
  - 077, Charlotte, North Carolina
  - 559, Charlotte, North Carolina
  - 058, Durham, North Carolina
  - 075, Wilmington, North Carolina
  - 061, Columbus, Ohio
  - 071, Middleburg Heights, Ohio
  - 041, Oklahoma City, Oklahoma
  - 076, Oklahoma City, Oklahoma
  - 097, Oklahoma City, Oklahoma
  - 547, Tulsa, Oklahoma
  - 032, Duncansville, Pennsylvania
  - 093, Philadelphia, Pennsylvania
  - 073, Pittsburgh, Pennsylvania
  - 094, Pittsburgh, Pennsylvania
  - 535, Charleston, South Carolina
  - 598, Myrtle Beach, South Carolina
  - 571, Jackson, Tennessee
  - 057, Memphis, Tennessee
  - 574, Amarillo, Texas
  - 078, Austin, Texas
  - 098, Austin, Texas
  - 570, Austin, Texas
  - 079, Dallas, Texas
  - 541, Houston, Texas
  - 563, Houston, Texas
  - 036, Mesquite, Texas
  - 066, San Antonio, Texas
  - 562, San Antonio, Texas
  - 534, Seattle, Washington
- Australia (5):
  - 429, Camperdown
  - 427, Clayton
  - 430, Liverpool
  - 425, Malvern
  - 426, Maroochydore
- Belgium (4):
  - 106, Brussels
  - 107, Brussels
  - 105, Leuven
  - 104, Liège
- Brazil (10):
  - 954, Belo Horizonte
  - 956, Campinas
  - 955, Goiânia
  - 950, Juiz de Fora
  - 453, Porto Alegre
  - 451, Recife
  - 450, Rio de Janeiro
  - 952, Rio de Janeiro
  - 452, Salvador
  - 454, São Paulo
- Bulgaria (5):
  - 200, Sofia
  - 202, Sofia
  - 203, Sofia
  - 204, Sofia
  - 205, Sofia
- Canada (6):
  - 500, London, Ontario
  - 502, Hamilton
  - 507, Mississauga
  - 508, Rimouski
  - 506, St. John's
  - 504, Toronto
- Czechia (3):
  - 218, Olomouc
  - 216, Prague
  - 215, Zlín
- 226, Tallinn, Estonia
- France (6):
  - 113, Lille
  - 618, Limoges
  - 617, Montpellier
  - 614, Paris
  - 116, Pessac
  - 616, Toulouse
- Germany (14):
  - 127, Berlin
  - 628, Berlin
  - 633, Berlin
  - 625, Cologne
  - 128, Frankfurt
  - 126, Freiburg im Breisgau
  - 637, Hamburg
  - 632, Herne
  - 626, Leipzig
  - 634, Mainz
  - 627, Münster
  - 129, Plochingen
  - 636, Roßlau
  - 631, Zerbst
- 349, Shatin, Hong Kong
- Hungary (7):
  - 712, Budapest
  - 716, Budapest
  - 718, Budapest
  - 717, Debrecen
  - 711, Szeged
  - 715, Szeged
  - 713, Zalaegerszeg
- Israel (9):
  - 378, Ashkelon
  - 376, Beersheba
  - 375, Haifa
  - 377, Haifa
  - 381, Jerusalem
  - 382, Kfar Saba
  - 380, Rehovot
  - 379, Tel Aviv
  - 383, Tel Litwinsky
- Italy (6):
  - 149, Ferrara
  - 648, Milan
  - 148, Padua
  - 647, Pisa
  - 646, Roma
  - 147, Torino
- Lithuania (3):
  - 242, Kaunas
  - 244, Klaipėda
  - 243, Vilnius
- Mexico (5):
  - 478, Guadalajara
  - 976, Mexico City
  - 982, Mexico City
  - 480, Mérida
  - 981, Torreón
- Poland (11):
  - 743, Bydgoszcz
  - 744, Częstochowa
  - 752, Elblag
  - 754, Elblag
  - 746, Katowice
  - 748, Lublin
  - 750, Lublin
  - 742, Poznan
  - 747, Szczecin
  - 751, Ustroń
  - 749, Warsaw
- Romania (10):
  - 263, Brasov
  - 260, Bucharest
  - 262, Bucharest
  - 264, Bucharest
  - 757, Bucharest
  - 758, Bucharest
  - 261, Cluj-Napoca
  - 759, Constanța
  - 756, Galati
  - 761, Iași
- Russia (4):
  - 779, Moscow
  - 285, Petrozavodsk
  - 284, Saint Petersburg
  - 281, Yekaterinburg
- South Africa (3):
  - 901, Cape Town
  - 902, Durban
  - 903, Stellenbosch
- South Korea (6):
  - 306, Busan
  - 303, Daegu
  - 308, Daejeon
  - 301, Incheon
  - 307, Seoul
  - 302, Suwon
- Spain (14):
  - 161, Barcelona
  - 661, Barcelona
  - 164, Bilbao
  - 660, Getafe
  - 662, Las Palmas de Gran Canaria
  - 162, Madrid
  - 163, Madrid
  - 664, Madrid
  - 166, Málaga
  - 165, San Cristóbal de La Laguna
  - 177, Santander
  - 663, Santiago de Compostela
  - 160, Seville
  - 659, Vigo
- Taiwan (4):
  - 325, Changhua
  - 326, Chiayi City
  - 328, Kaohsiung City
  - 330, Taipei
- Ukraine (8):
  - 791, Donetsk
  - 799, Ivano-Frankivsk
  - 790, Kiev
  - 794, Kiev
  - 797, Kiev
  - 792, Luhansk
  - 793, Odesa
  - 796, Vinnytsia
- United Kingdom (5):
  - 677, Birmingham
  - 178, Brighton
  - 182, Doncaster
  - 179, Leeds
  - 181, Romford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in July 2011 and concluded in February 2016.
Pre-assignment Details: Participant Flow refers to the Enrolled Set, that consisted of all subjects who gave informed consent.
Groups:
- Enrollment Cohort 1 Epratuzumab 600 mg Per Week (ES): Enrolled Set (ES) of subjects enrolled prior to the approval of Protocol Amendment 2. 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
- Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (ES): Enrolled Set (ES) of subjects enrolled prior to the approval of Protocol Amendment 2
  1200 mg infusions delivered every other week (Q2W) for a total of 4 weeks (cumulative dose 2400 mg) over sixteen 12 week treatment cycles
- Enrollment Cohort 2 Epratuzumab 600 mg Per Week (ES): Enrolled Set (ES) of subjects enrolled prior to the approval of Protocol Amendment 2
  600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
Period: Overall Study
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (ES) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (ES) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (ES)
Started | 244 | 498 | 508
Completed | 56 | 0 | 0
Not Completed | 188 | 498 | 508
Not completed — Lack of Efficacy | 17 | 30 | 48
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Lost to Follow-up | 10 | 9 | 17
Not completed — Withdrawal by Subject | 34 | 60 | 66
Not completed — Sponsor terminated study | 89 | 333 | 330
Not completed — AE, serious fatal | 4 | 4 | 1
Not completed — SAE, non-fatal | 11 | 23 | 14
Not completed — AE, non-serious non-fatal | 12 | 19 | 11
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 0 | 1 | 1
Not completed — AE, unknown type | 0 | 1 | 0
Not completed — Other | 10 | 16 | 18

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Enrolled Set, that consisted of all subjects who gave informed consent.
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (ES) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (ES) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (ES) | Total Title
Number analyzed (Participants) | 244 | 498 | 508 | 1250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 239 | 489 | 490 | 1218
  >=65 years | 5 | 9 | 18 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.0) | 41.9 (11.5) | 42.5 (11.9) | 42.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 467 | 478 | 1171
  Male | 18 | 31 | 30 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Prematurely Discontinuing Due to a Treatment-emergent Adverse Event (TEAE) During the Treatment Period (Maximum 96 Weeks)
Description: A TEAE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Time Frame: During the treatment period (through Week 96)
Population: Safety Set (SS) which consisted of all subjects who had received at least 1 partial dose of study medication during SL0012. A partial dose of study medication was defined as any infusion during which the subject received more than (>) 0mL of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- All Epratuzumab 600 mg Per Week: 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
- All Subjects: Subjects receiving 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles and subjects receiving 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over sixteen 12 week treatment cycles
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (ES) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (ES) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (ES) | All Epratuzumab 600 mg Per Week | All Subjects
Number analyzed (Participants) | 244 | 497 | 507 | 751 | 1248
Participants | 26 | 45 | 25 | 51 | 96

2. Primary Outcome: Percentage of Subjects Prematurely Discontinuing Due to a Treatment-emergent Adverse Event (TEAE) During the Treatment Period (Maximum 96 Weeks)
Description: as for outcome 1
Time Frame: During the treatment period (through Week 96)
Population: Safety Set (SS) which consisted of all subjects who had received at least 1 partial dose of study medication during SL0012. A partial dose of study medication was defined as any infusion during which the subject received >0mL of study medication.
Measure: Number; unit: percentage of participants
Groups:
- Enrollment Cohort 1 Epratuzumab 600 mg Per Week: Subjects enrolled prior to the approval of Protocol Amendment 2. 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
- Enrollment Cohort 2 Epratuzumab 1200 mg Q2W: Subjects enrolled after approval of Protocol Amendment 2. 1200 mg infusions delivered every other week (Q2W) for a total of 4 weeks (cumulative dose 2400 mg) over sixteen 12 week treatment cycles
- Enrollment Cohort 2 Epratuzumab 600 mg Per Week: Subjects enrolled after approval of Protocol Amendment 2. 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W | Enrollment Cohort 2 Epratuzumab 600 mg Per Week | All Epratuzumab 600 mg Per Week | All Subjects
Number analyzed (Participants) | 244 | 497 | 507 | 751 | 1248
percentage of participants | 10.7 | 9.1 | 4.9 | 6.8 | 7.7

3. Primary Outcome: Number of Subjects Reporting at Least 1 Serious Adverse Event (SAE) During the Treatment Period (Maximum 96 Weeks)
Description: A SAE is a treatment-emergent adverse event (TEAE) that the investigator classifies as serious. This includes:
  * Death
  * Life-threatening
  * Significant or persistent disability/incapacity
  * Congenital anomaly/birth defect (including that occurring in a fetus)
  * Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious
  * Initial inpatient hospitalization or prolongation of hospitalization
Time Frame: During the treatment period (through Week 96)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W | Enrollment Cohort 2 Epratuzumab 600 mg Per Week | All Epratuzumab 600 mg Per Week | All Subjects
Number analyzed (Participants) | 244 | 497 | 507 | 751 | 1248
Participants | 81 | 119 | 104 | 185 | 304

4. Primary Outcome: Percentage of Subjects Reporting at Least 1 Serious Adverse Event (SAE) During the Treatment Period (Maximum 96 Weeks)
Description: as for outcome 3
Time Frame: During the treatment period (through Week 96)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W | Enrollment Cohort 2 Epratuzumab 600 mg Per Week | All Epratuzumab 600 mg Per Week | All Subjects
Number analyzed (Participants) | 244 | 497 | 507 | 751 | 1248
percentage of participants | 33.2 | 23.9 | 20.5 | 24.6 | 24.4

5. Secondary Outcome: Number of Subjects Meeting Treatment Response Criteria According to a Combined Response Index
Description: Combined response index is a response variable (yes/no) incorporating the following criteria for achievement of responder status (ie, all criteria must be met to achieve responder status): (1) British Isles Lupus Activity Group (BILAG) improvement, (2) No worsening in Systemic Lupus Erythematosus Activity Index (SLEDAI), (3) No worsening in Physician's Global Assessment of Disease, and (4) No disallowed changes in concomitant medications, with disallowed changes including mainly increases in corticosteroids, immunosuppressants, and antimalarials.
Time Frame: At Week 48
Population: The Full Analysis Subset 1 (FASS1) consisted of all subjects in the FAS who were enrolled in study SL0008 (NCT00660881), SL0009 (NCT01262365) or SL0010 (NCT01261793) prior to enrollment in SL0012.
Measure: Count of Participants; unit: Participants
Groups:
- Enrollment Cohort 1 Epratuzumab 600 mg Per Week (FASS1); Enrollment Cohort 2 Epratuzumab 600 mg Per Week (FASS1); All Epratuzumab 600 mg Per Week (FASS1): Full Analysis Subset 1 (FASS1) consisted of all subjects in the FAS who were enrolled in study SL0008 (NCT00660881), SL0009 (NCT01262365), or SL0010 (NCT01261793) prior to enrollment in SL0012.
  Subjects were enrolled prior to the approval of Protocol Amendment 2. 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles
- Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (FASS1): Full Analysis Subset 1 (FASS1) consisted of all subjects in the FAS who were enrolled in study SL0008 (NCT00660881), SL0009 (NCT01262365), or SL0010 (NCT01261793) prior to enrollment in SL0012.
  Subjects were enrolled prior to the approval of Protocol Amendment 2. 1200 mg infusions delivered every other week (Q2W) for a total of 4 weeks (cumulative dose 2400 mg) over sixteen 12 week treatment cycles
- All Subjects (FASS1): Full Analysis Subset 1 (FASS1) consisted of all subjects in the FAS who were enrolled in study SL0008 (NCT00660881), SL0009 (NCT01262365), or SL0010 (NCT01261793) prior to enrollment in SL0012.
  Subjects were enrolled prior to the approval of Protocol Amendment 2. Subjects receiving 600 mg infusions delivered weekly for a total of 4 consecutive weeks (cumulative dose 2400 mg) over sixteen 12-week treatment cycles and subjects receiving 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over sixteen 12 week treatment cycles
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (FASS1) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (FASS1) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (FASS1) | All Epratuzumab 600 mg Per Week (FASS1) | All Subjects (FASS1)
Number analyzed (Participants) | 230 | 488 | 494 | 724 | 1212
Participants | 82 | 146 | 134 | 216 | 362

6. Secondary Outcome: Percentage of Subjects Meeting Treatment Response Criteria According to a Combined Response Index
Description: as for outcome 5
Time Frame: Week 48
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (FASS1) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (FASS1) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (FASS1) | All Epratuzumab 600 mg Per Week (FASS1) | All Subjects (FASS1)
Number analyzed (Participants) | 230 | 488 | 494 | 724 | 1212
percentage of participants | 35.7 | 29.9 | 27.1 | 29.8 | 29.9

7. Secondary Outcome: Number of Subjects Meeting Treatment Response Criteria According to a Combined Response Index
Description: as for outcome 5
Time Frame: Week 96
Population: The Full Analysis Subset 1 (FASS1) consisted of all subjects in the FAS who were enrolled in study SL0008 (NCT00660881), SL0009 (NCT01262365) or SL0010 (NCT01261793) prior to enrollment in SL0012, and with available results at the Week 96 time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (FASS1) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (FASS1) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (FASS1) | All Epratuzumab 600 mg Per Week (FASS1) | All Subjects (FASS1)
Number analyzed (Participants) | 186 | 306 | 298 | 484 | 790
Participants | 74 | 66 | 78 | 152 | 218

8. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria According to a Combined Response Index
Description: as for outcome 5
Time Frame: Week 96
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (FASS1) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (FASS1) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (FASS1) | All Epratuzumab 600 mg Per Week (FASS1) | All Subjects (FASS1)
Number analyzed (Participants) | 186 | 306 | 298 | 484 | 790
percentage of participants | 39.8 | 21.6 | 26.2 | 31.4 | 27.6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 1 until Safety Follow-Up Visit (up to Week 196)
Arm/Group | Enrollment Cohort 1 Epratuzumab 600 mg Per Week | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W | Enrollment Cohort 2 Epratuzumab 600 mg Per Week | All Epratuzumab 600 mg Per Week | All Subjects
All-Cause Mortality (participants affected / at risk) | 4/244 | 4/497 | 1/507 | 5/751 | 9/1248
Serious Adverse Events (participants affected / at risk) | 81/244 | 119/497 | 104/507 | 185/751 | 304/1248
Other Adverse Events (participants affected / at risk) | 177/244 | 296/497 | 306/507 | 483/751 | 779/1248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (N=244) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (N=497) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (N=507) | All Epratuzumab 600 mg Per Week (N=751) | All Subjects (N=1248)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (3) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Splenic cyst (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleuropericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinoatrial block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Factor VII deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Necrotising retinitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Panophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retinal disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (3) | 3 (3) | 4 (5) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 3 (4) | 4 (5)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 1 (3) | 2 (4)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Oesophageal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 4 (4) | 8 (9) | 9 (10) | 13 (14)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Drug interaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Local swelling (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Serositis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (3)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis migration (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 7 (7) | 9 (10) | 15 (16) | 22 (23)
Sepsis (Infections and infestations) | 3 (4) | 3 (3) | 4 (4) | 7 (8) | 10 (11)
Cellulitis (Infections and infestations) | 1 (1) | 4 (4) | 3 (5) | 4 (6) | 8 (10)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 7 (7)
Arthritis bacterial (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 3 (4)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 3 (4)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Meningitis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 3 (4)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Biopsy liver (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood cortisol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (15) | 12 (12) | 19 (19) | 32 (34)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 2 (2) | 3 (3) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (5) | 4 (5) | 6 (7)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 6 (6) | 6 (6)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 4 (4)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (2) | 3 (4)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 2 (3)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lupus encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropsychiatric lupus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Seizure anoxic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thecal sac compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 6 (6)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 3 (4)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kidney fibrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 4 (4)
Endometriosis (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Polymedication (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Venous thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrollment Cohort 1 Epratuzumab 600 mg Per Week (N=244) | Enrollment Cohort 2 Epratuzumab 1200 mg Q2W (N=497) | Enrollment Cohort 2 Epratuzumab 600 mg Per Week (N=507) | All Epratuzumab 600 mg Per Week (N=751) | All Subjects (N=1248)
Nausea (Gastrointestinal disorders) | 39 (80) | 59 (86) | 62 (79) | 101 (159) | 160 (245)
Diarrhoea (Gastrointestinal disorders) | 27 (41) | 47 (58) | 34 (47) | 61 (88) | 108 (146)
Vomiting (Gastrointestinal disorders) | 22 (45) | 32 (43) | 29 (38) | 51 (83) | 83 (126)
Fatigue (Gastrointestinal disorders) | 17 (24) | 19 (22) | 21 (22) | 38 (46) | 57 (68)
Upper respiratory tract infection (Infections and infestations) | 66 (140) | 76 (126) | 82 (120) | 148 (260) | 224 (386)
Urinary tract infection (Infections and infestations) | 56 (124) | 61 (88) | 62 (90) | 118 (214) | 179 (302)
Nasopharyngitis (Infections and infestations) | 38 (56) | 42 (65) | 45 (67) | 83 (123) | 125 (188)
Bronchitis (Infections and infestations) | 34 (38) | 35 (38) | 35 (41) | 69 (79) | 104 (117)
Sinusitis (Infections and infestations) | 25 (40) | 41 (48) | 38 (48) | 63 (88) | 104 (136)
Influenza (Infections and infestations) | 15 (16) | 22 (24) | 21 (23) | 36 (39) | 58 (63)
Gastroenteritis (Infections and infestations) | 14 (14) | 19 (21) | 17 (23) | 31 (37) | 50 (58)
Conjunctivitis (Infections and infestations) | 14 (16) | 15 (17) | 8 (8) | 22 (24) | 37 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (47) | 31 (32) | 32 (32) | 66 (79) | 97 (111)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (40) | 36 (44) | 30 (38) | 54 (78) | 90 (122)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 15 (19) | 18 (26) | 23 (30) | 38 (49) | 56 (75)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (21) | 15 (17) | 19 (21) | 34 (42) | 49 (59)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 (14) | 18 (20) | 6 (7) | 19 (21) | 37 (41)
Bursitis (Musculoskeletal and connective tissue disorders) | 15 (24) | 9 (11) | 7 (7) | 22 (31) | 31 (42)
Headache (Nervous system disorders) | 46 (66) | 67 (84) | 57 (80) | 103 (146) | 170 (230)
Dizziness (Nervous system disorders) | 20 (26) | 23 (30) | 23 (25) | 43 (51) | 66 (81)
Hypoaesthesia (Nervous system disorders) | 13 (15) | 9 (9) | 12 (13) | 25 (28) | 34 (37)
Depression (Psychiatric disorders) | 16 (17) | 23 (23) | 15 (16) | 31 (33) | 54 (56)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (25) | 30 (31) | 32 (43) | 53 (68) | 83 (99)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 (24) | 9 (11) | 14 (16) | 29 (40) | 38 (51)
Urticaria (Respiratory, thoracic and mediastinal disorders) | 13 (20) | 7 (7) | 4 (4) | 17 (24) | 24 (31)
Hypertension (Vascular disorders) | 17 (19) | 26 (28) | 26 (27) | 43 (46) | 69 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days